CLINICAL TRIAL: NCT03179592
Title: VOLtage-based Contrast Media AdaptatioN in Coronary Computed Tomography Angiography (VOLCANIC-CTA): A Prospective Trial
Brief Title: VOLtage-based Contrast Media AdaptatioN in Coronary Computed Tomography Angiography
Acronym: VOLCANIC-CTA
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00060805
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases
Keywords: Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — iopromide; Injections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Low-volume contrast media injection protocol: Patients will receive a low-volume contrast media (Ultravist 370Mg I/Ml Solution for Injection) injection protocol that is tailored to a specific tube voltage. Tube voltages will be automatically selected by the scanner to be used for the CCTA acquisition.
  Interventions: Drug: Ultravist 370Mg I/Ml Solution for Injection

INTERVENTIONS:
Drug: Ultravist 370Mg I/Ml Solution for Injection — Reduced contrast-volume injection protocols based on patient specific tube voltage.
  Other Names: Iopromide

SUMMARY:
The purpose of this study is to prospectively evaluate the effectiveness of low-volume contrast media (CM) injection protocols adapted to tube voltage in patients undergoing Coronary Computed Tomography Angiography (CCTA).

ELIGIBILITY:
Inclusion Criteria:

1. Referred for a clinically indicated CCTA scan.
2. Subject must be 18 - 85 years of age.
3. Subject must provide written informed consent prior to any study-related procedures being performed.
4. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

1. Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

   * By testing (serum or urine beta HCG) within 24 hours before study agent administration, or
   * By surgical sterilization, or
   * Post-menopausal, with minimum one (1) year history without menses.
2. Subject is chosen by the automated tube voltage selection algorithm (or adjusted by the technologist) to be scanned using a tube voltage that is not 70, 80, 90, 100, 110, 120, or 130 kV.
3. Subject is chosen by the automated tube voltage selection algorithm (or adjusted by the technologist) to be scanned using a tube voltage that has previously reached the maximum subject number (20 subjects per tube voltage).
4. Subject has an acute psychiatric disorder.
5. Subject is unwilling to comply with the requirements of the protocol.
6. Subject has previously entered this study.
7. Subject has an allergy against iodinated contrast agents or pharmaceutical stressors used in this study.
8. Subject has impaired renal function (creatinine > 1.5 mg/dl).
9. Subject is in unstable condition.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes 120 patients who present to radiology department for clinically indicated CCTA scan. In order to be included patients must meet all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of image quality | 2 years
  This will be performed by two independent observers using a semi-quantitative rating scale of 1 - 5. Image quality will be graded on a five-point scoring system: 1 non-diagnostic; 2 limited diagnostic value; 3 adequate (presence of artifacts not limiting detection of luminal stenosis); 4 good; 5 excellent. Image quality assessments will be performed on both the investigative and control groups.
Quantitative assessment of image quality | 2 years
  Measurements and calculations will be performed by two independent observers who will be blinded to image acquisition parameters. Signal-to-noise ratio (SNR) and contrast-to-noise ratio (CNR) will be measured for all images.

SECONDARY OUTCOMES:
Radiation dose of coronary CTA | 2 years
  Determine the radiation dose (mSv) associated with low-volume contrast injection CCTA protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No